CLINICAL TRIAL: NCT00901485
Title: Autotitrating Non-invasive Ventilation (NIV) Versus Standard NIV; a Randomised Crossover Trial in Patients With Newly Diagnosed Hypoventilation
Brief Title: Autotitrating Versus Standard Non-invasive Ventilation (NIV) in Newly Diagnosed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 08/H0708/16; R&D No. 2008/LF017B (Other: Research & Development Department, RBH)
Record Dates: First submitted 2009-01-14; First posted 2009-05-13 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Nocturnal Hypoventilation; Neuromuscular Disease; Chest Wall Disorder
Keywords: Respiratory insufficiency; Hypercapnia; Hypoventilation; Sleep; Polysomnography; Hypoxia; Titration; Non Invasive Ventilation
MeSH Terms: conditions — Neuromuscular Diseases; Respiratory Insufficiency; Hypercapnia; Hypoventilation; Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- autotitrating NIV (Experimental): approximately 6 weeks using domiciliary nocturnal autotitrating non-invasive ventilation
  Interventions: Device: AutoVPAP
- Standard non-invasive ventilation (Active Comparator): approximately 6 weeks using domiciliary nocturnal standard non-invasive ventilation
  Interventions: Device: VPAPIIIST-A

INTERVENTIONS:
Device: AutoVPAP — Automatically titrated non-invasive ventilator, with target gross alveolar ventilation and back up respiratory rate determined by learn function. Nocturnal use for one month in patient's home.
  Other Names: autotitrating variable positive airway pressure; autotitrating NIV; automatically titrating NIV
  Arms: autotitrating NIV
Device: VPAPIIIST-A — Standard non-invasive ventilator with pressure and respiratory rate settings determined by healthcare professional. Nocturnal use for one month in the patient's home.
  Other Names: standard NIV; standard non-invasive ventilator; variable positive airway pressure; VPAP
  Arms: Standard non-invasive ventilation

SUMMARY:
The aim of the study is to compare the efficacy and tolerance of autotitrating non-invasive ventilation (NIV) versus standard NIV in patients with newly diagnosed nocturnal hypoventilation who have never experienced nocturnal, home NIV.

DETAILED DESCRIPTION:
The aim of the study is to compare the effect of two types of noninvasive ventilator (a small machine that assists breathing) in patients newly diagnosed with nocturnal hypoventilation who are inexperienced in the use of noninvasive ventilation (NIV). NIV is standard therapy for patients with nocturnal hypoventilation.

The most common type of NIV is bilevel pressure support which assists patient breathing by delivering different levels of air pressure during inspiration and expiration via a mask covering the nose or nose and mouth. Standard bilevel NIV (VPAP™) has been further developed to create a new automatically adjusting NIV (AutoVPAP™). Automatically adjusting NIV varies the inspiratory air pressure according to the airflow rates generated by the patient. This may improve patient comfort, hours of NIV use and recovery time.

Patients over the age of 18 referred to, or under follow up at, the Royal Brompton Hospital who require domiciliary NIV but are inexperienced with use of NIV will be considered for entry into this randomised crossover study. If eligible for inclusion and willing to take part patients will be setup on automatically adjusting NIV or standard NIV, assigned in random order. At the end of one month the patient will be swapped to the alternative NIV for a further one month of domiciliary NIV treatment. At the end of each one month treatment period the patient will undergo overnight polysomnography, transcutaneous CO2 monitoring and 24 hour Holter monitoring.

ELIGIBILITY:
Inclusion Criteria:

* new clinical diagnosis of nocturnal hypoventilation
* requirement for long-term domiciliary non-invasive ventilation
* no previous experience with domiciliary non-invasive ventilation

Exclusion Criteria:

* uncontrolled cardiac failure
* acute exacerbation of respiratory failure
* daytime resting PaO2 < 7.5kPa
* moderate or severe bulbar weakness
* inability to understand rationale and/or consent form for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Simonds, MD, FRCP, Principal Investigator — Royal Brompton & Harefield Hospital NHS Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- AutoVPAP Then VPAPIIIST-A; VPAPIIIST-A First, Then AutoVPAP: All patients underwent a cross over design -
  1 month using domiciliary nocturnal standard non-invasive ventilation. (VPAPIIIST-A), and one month using AutoTitrating non-invasive ventilation
Period: Overall Study
Arm/Group | AutoVPAP Then VPAPIIIST-A | VPAPIIIST-A First, Then AutoVPAP
Started | 10 | 13
Completed | 9 | 9
Not Completed | 1 | 4
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Patients underwent a cross over study design. In a randomised order they used 1 month of domiciliary nocturnal autotitrating, intelligent volume assured pressure support (iVAPS) non-invasive ventilation, and one month of standard non-invasive ventilation
Arm/Group | All Patients
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 54 [43 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
FEV1 (forced expiratory volume) (L) [Median (Inter-Quartile Range); unit: L] | 1.5 [0.8 to 1.9]
FVC (forced vital capacity) [Median (Inter-Quartile Range); unit: L] | 1.9 [1.4 to 2.7]
FEV1/FVC [Median (Inter-Quartile Range); unit: ratio] | 0.75 [0.64 to 0.82]
maximal inspiratory effort (MIP) (cmH2O) [Median (Inter-Quartile Range); unit: cmH2O] | 50 [30 to 72]
Maximum expiratory pressure (MEP) [Median (Inter-Quartile Range); unit: cmH2O] | 118 [59 to 143]
sniff nasal inspiratory pressure (SNIP) [Median (Inter-Quartile Range); unit: cmH2O] | 39 [23 to 56]

OUTCOME MEASURES:

1. Primary Outcome: Overnight Mean Oxygen Saturation
Description: Overnight oximetry (SaO2) and transcutaneous capnography (PtcCO2) (TOSCA, Linde Medical Sensors, Switzerland) were performed during a sleep a on NIV at the end of each month's NIV therapy.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: % SaO2
Groups:
- Autotitrating iVAPS NIV: AutoVPAP: Automatically titrated non-invasive ventilator, with target gross alveolar ventilation and back up respiratory rate determined by learn function. Nocturnal use for one month in patient's home.
  All completing patients used iVAPS in either period1 or period 2. The results are for all patients after the 1 month of iVAPS NIV therapy.
- Standard Non-invasive PS Ventilation: VPAPIIIST-A: Standard non-invasive ventilator with pressure and respiratory rate settings determined by healthcare professional. Nocturnal use for one month in the patient's home.
  All completing patients used iVAPS in either period1 or period 2. The results are for all patients after the 1 month of standard PS NIV therapy.
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 18 | 18
% SaO2 | 96 [95 to 98] | 96 [93 to 97]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; We tested the hypothesis that iVAPS can ventilate a patient naive to NIV at least as effectively as standard PS. Sleep and breathing parameters at the end of each treatment period were compared using Wilcoxon Signed Rank test. The median difference between treatments with 95% confidence intervals was then compared by related-samples Hodges-Lehman test; Test type: Non-Inferiority or Equivalence — To test for non-inferiority, a sample size of 36 (18 patients completing both arms of the crossover) was calculated to provide 80% power to detect a 2.5% drop in the primary outcome, mean overnight oxygen saturation (SpO2), with a SD of 3% at a significance level of 0.05; p = 0.13, Wilcoxon (Mann-Whitney) — a priori threshold for significance p<0.05; Median Difference (Final Values) = 0.4, 95% CI 2-sided [-0.2 to 1.0]

2. Secondary Outcome: Overnight Mean Transcutaneous Carbon Dioxide
Description: as for outcome 1
Time Frame: 4 weeks
Population: All patients had a sleep study after 1 month of each mode of ventilation and all results are included in this analysis
Measure: Median (Inter-Quartile Range); unit: kPa
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 18 | 18
kPa | 6.5 [5.8 to 6.8] | 6.2 [5.8 to 6.9]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Hypothesis: that we tested the hypothesis that iVAPS, with automated selection of ventilator settings, was non-inferior to standard pressure support (PS) ventilation, with settings determined by an experienced healthcare professional, for controlling nocturnal hypoventilation in patients naïve to NIV; Test type: Non-Inferiority or Equivalence — PtcCO2 is compared as a secondary outcome resulting in CO2 elimination similar to that of standard PS ventilation (median difference (95% CI) of -0.04(- 0.03 to 0.4)kPa in mean overnight PtcCO2); p = 0.54, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-0.3 to 0.4]

3. Secondary Outcome: Overnight Peak Transcutaneous Carbon Dioxide
Description: as for outcome 1
Time Frame: 4 weeks
Population: All patients had a sleep study after 1 month of each mode of ventilation and all results are included in this analysis
Measure: Median (Inter-Quartile Range); unit: kPa
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 18 | 18
kPa | 7.1 [6.3 to 7.6] | 6.9 [6.3 to 7.5]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.94, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0, 95% CI 2-sided [-0.5 to 0.5]

4. Secondary Outcome: Oxygen Desaturation Index (>4%)
Description: Overnight oximetry (SaO2) and transcutaneous capnography (PtcCO2) (TOSCA, Linde Medical Sensors, Switzerland) were performed during a sleep a on NIV at the end of each month's NIV therapy. ODI is the number of events per hour that SaO2 drops by >4%.
Time Frame: 4 weeks
Population: All patients had a sleep study after 1 month of each mode of ventilation and all results are included in this analysis
Measure: Median (Inter-Quartile Range); unit: events/hr
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 18 | 18
events/hr | 2.5 [1.3 to 12.2] | 5.0 [1.5 to 11.6]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.42, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1, 95% CI 2-sided [-2 to 1]

5. Secondary Outcome: Sleep Quality: Arousal Index
Description: A full PSG was performed during a sleep a on NIV at the end of each month's NIV therapy. Standard polysomnography analysis was performed by two team members blinded to patient identity and ventilator mode (REP/JJ).
  Sleep quality was assessed by the Arousal Index (no of arousals/hour)
Time Frame: 4 weeks
Population: 16 patients had comparative PSG data with all signals present for their sleep studies on both ventilator modes.
Measure: Median (Inter-Quartile Range); unit: events/hour
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 16 | 16
events/hour | 17 [8 to 24] | 14 [10 to 26]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.82, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0, 95% CI [-8 to 4]

6. Other Pre Specified Outcome: Ventilator Adherence
Description: Summary data from the ventilators were downloaded after each month's therapy, including adherence (hours of use), and ventilator output (nightly mean pressure support, minute ventilation (MV), RR and leak).
Time Frame: 4 weeks
Population: 1 participant had missing adherence data and so was excluded from this analysis
Measure: Median (Inter-Quartile Range); unit: hh:mm/day
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 17 | 17
hh:mm/day | 5.40 [4.42 to 6.49] | 4.20 [2.27 to 6.17]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.0004, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1.04, 95% CI 2-sided [0.27 to 1.44]

7. Other Pre Specified Outcome: Median Overnight Minute Ventilation
Description: as for outcome 6
Time Frame: 4 weeks
Population: 2 patients had missing values from one of the ventilator modes, thus were excluded from the analysis
Measure: Median (Inter-Quartile Range); unit: L/min
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 16 | 16
L/min | 6.8 [5.3 to 8.3] | 6.2 [5.4 to 9.4]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.5, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.2 to 0.5]

8. Other Pre Specified Outcome: Median Overnight Pressure Support
Description: as for outcome 6
Time Frame: 4 weeks
Population: 2 patients had missing data from one of the ventialtory modes and were excluded from the analysis
Measure: Median (Inter-Quartile Range); unit: cmH2O
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 16 | 16
cmH2O | 8.3 [5.6 to 10.4] | 10.0 [9.0 to 11.4]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.001, Wilcoxon (Mann-Whitney); Median Difference (Net) = -2.2, 95% CI 2-sided [-4.5 to 0.3]

9. Other Pre Specified Outcome: Median Overnight Tidal Volume
Description: as for outcome 6
Time Frame: 4 weeks
Population: 2 patients had missing data from one of the ventilatory modes and so were excluded
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 16 | 16
ml | 421 [321 to 521] | 400 [300 to 575]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.47, Wilcoxon (Mann-Whitney); Median Difference (Net) = -10, 95% CI 2-sided [-54 to 23]

10. Other Pre Specified Outcome: Median Overnight Respiratory Rated
Description: as for outcome 6
Time Frame: 4 weeks
Population: 2 patients had missing data from one ventilatory mode and thus were excluded from analysis
Measure: Median (Inter-Quartile Range); unit: bpm
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 16 | 16
bpm | 16.7 [13.2 to 18.4] | 15.5 [13.5 to 17.0]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.41, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.3, 95% CI 2-sided [-0.7 to 2.2]

11. Other Pre Specified Outcome: Subjective Ventilator Tolerance: Comfort of Breath Delivered
Description: Subjective tolerance of ventilator modes was assessed by 10cm visual analogue scales (VAS) in response to questions on comfort of breath, ease of falling asleep, use of ventilator, and mode preference. VAS was scored from 0-100 for each question (0 - negative and 100 -s positive)
Time Frame: 4 weeks
Population: 2 patients had missing data and thus were excluded from analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 16 | 16
units on a scale | 73 [55 to 91] | 72 [45 to 85]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.36, Wilcoxon (Mann-Whitney); Median Difference (Net) = 4, 95% CI 2-sided [-5 to 12]

12. Other Pre Specified Outcome: Subjective Ventilator Tolerance: Ease of Falling Asleep
Description: as for outcome 11
Time Frame: 4 weeks
Population: 2 patients had missing data and so were excluded from analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 16 | 16
units on a scale | 86 [69 to 94] | 79 [60 to 89]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.59, Wilcoxon (Mann-Whitney); Median Difference (Net) = 2, 95% CI 2-sided [-5 to 14]

13. Other Pre Specified Outcome: Subjective Ventilation Tolerance: Ease of Use of Ventilator
Description: as for outcome 11
Time Frame: 4 weeks
Population: 2 patients had missing data and were thus excluded from analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 16 | 16
units on a scale | 90 [77 to 95] | 86 [78 to 98]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.59, Wilcoxon (Mann-Whitney); Median Difference (Net) = 2, 95% CI 2-sided [-5 to 14]

14. Other Pre Specified Outcome: Subjective Ventilator Tolerance: Liked Using Ventilator
Description: as for outcome 11
Time Frame: 4 weeks
Population: 2 patients had missing data, thus were excluded from analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
Number analyzed (Participants) | 16 | 16
units on a scale | 81 [55 to 94] | 68 [24 to 79]
Statistical Analysis 1: Comparison: Autotitrating iVAPS NIV vs Standard Non-invasive PS Ventilation; Test type: Non-Inferiority or Equivalence — This is a secondary outcome; p = 0.72, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1, 95% CI 2-sided [-9 to 5]

15. Other Pre Specified Outcome: Ventilator Mode Preference
Description: as for outcome 11
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the entire course of the trial; each participant was monitored throughout their participation of 2 months (1 month on each ventilator).
Arm/Group | Autotitrating iVAPS NIV | Standard Non-invasive PS Ventilation
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No